CLINICAL TRIAL: NCT06928090
Title: A Retrospective Observational Study of Efficacy and Safety of DTG/3TC(Dolutegravir/Lamivudine) in Treatment-naïve HIV-1 Infected Patients From at Real-life Cohort in Korea
Brief Title: Efficacy and Safety of DTG/3TC in Treatment-naïve HIV-1 Infected Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Chungnam National University Hospital (Other)
Responsible Party: Principal Investigator, Yeon-sook, Kim, Professor, Chungnam National University Hospital
Other Study IDs: CNUH 2024-10-046
Record Dates: First submitted 2025-03-27; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: HIV
MeSH Terms: interventions — dolutegravir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- DTG/3TC: Single arm cohort
  Interventions: Drug: DTG + 3TC FDC

INTERVENTIONS:
Drug: DTG + 3TC FDC — None(Non-interventional, retrospective chart review, single-arm study )

SUMMARY:
Non-interventional, retrospective, single arm study of individuals who have initiated a DTG/3TC regimen. Medical chart will be reviewed by the investigators. Naive subjects will be identified by the clinic database as having initiated DTG/3TC.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 diagnosis
* Prescribed DTG/3TC alone to manage HIV-1 infection as initial antiretroviral treatment at the study centers

Exclusion Criteria:

* HIV-2 diagnosis
* Previous antiretroviral treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Estimated enrollment: 150-200 subjects.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients achieving viral suppression | At week 48 after DTG/3TC treatment
  Virological suppression is HIV RNA viral load < 50 copies/mL

SECONDARY OUTCOMES:
Change in CD4+cell counts | From baseline to week 48
  Change in CD4+ T-cell count from baseline
Persistence on DTG/3TC | At 48 weeks
  The percentage of patients remaining on DTG/3TC over time after initiating DTG/3TC.
Reasons for Discontinuation | Up to 48 weeks.
  Reason for discontinuation (HBV co-infection, Virological Failure, Blip, Simplification, Drug-drug Interactions, AE/SAE, Pregnancy, Cost, Patient Preference, Follow-up loss))
Changes in BMI | From baseline to week 48
  Changes from baseline BMI( kg/m^2) in treatment-Naive
Changes of lipid profile | From baseline to week 48
  Changes of lipid profile from basliene in treatment-Naive. These changes include increased levels of total cholesterol, low-density lipoprotein cholesterol and high-density lipoprotein cholesterol, triglycerides.

CONTACTS AND LOCATIONS:
Overall Officials: Yeon-sook kim, Study Director — Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospital, 282 Munwha-ro, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: Undecided